CLINICAL TRIAL: NCT03660865
Title: A Prospective, Randomized, Controlled, Multi-center Clinical Study to Evaluate the Safety and Effectiveness of the RxSight Light Adjustable Lens (LAL) in Subjects With Prior Corneal Refractive Surgery
Brief Title: Clinical Study to Evaluate the Safety and Effectiveness of the RxSight Light Adjustable Lens (LAL) in Subjects With Prior Corneal Refractive Surgery
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: RxSight, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CSP-027
Record Dates: First submitted 2018-08-29; First posted 2018-09-07 (Actual); Results first posted 2021-11-22 (Actual); Last update posted 2021-12-23 (Actual); Status verified 2021-11

CONDITIONS: Aphakia; Cataract
Keywords: Light Adjustable Lens; Intraocular lens; LAL
MeSH Terms: conditions — Aphakia; Cataract

STUDY DESIGN:
Intervention Model Description: All subjects will receive the same treatment; however, each subject will have their eyes randomized to receive the experimental treatment in either the left/right eye. The control will then be assigned to the other.
Masking Description: Select post operative assessments will be performed on both the experimental and control eye by an examiner who will be masked to the eye assignments.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes

ARMS (2):
- Light adjustable lens (LAL) and Light Delivery Device (LDD) (Experimental): A pre-determined randomization scheme will be utilized to designate each of the patient's eyes as the primary eye (LAL) or the fellow eye (Control). Patient's primary eye will receive the light adjustable lens.
  Interventions: Device: Light Adjustable lens (LAL) and Light Delivery Device (LDD)
- Control IOL (Active Comparator): A pre-determined randomization scheme will be utilized to designate each of the patient's eyes as the primary eye (LAL) or the fellow eye (Control). Patient's fellow eye will receive the control IOL.
  Interventions: Device: Control IOL

INTERVENTIONS:
Device: Light Adjustable lens (LAL) and Light Delivery Device (LDD) — Primary eye will receive Light adjustable lens with Light delivery Device treatments
  Arms: Light adjustable lens (LAL) and Light Delivery Device (LDD)
Device: Control IOL — Fellow eye will receive control IOL
  Arms: Control IOL

SUMMARY:
The primary objective of this study is to evaluate, for the visual correction of aphakia, the safety and effectiveness of the RxSight Light Adjustable Lens (LAL) and Light Delivery Device (LDD) to reduce postoperative refractive error and improve uncorrected distance visual acuity in eyes with prior corneal refractive surgery. A control group consisting of fellow eyes implanted with a commercially available IOL will be used to compare the safety and effectiveness of the LAL.

ELIGIBILITY:
Inclusion Criteria:

* Must sign a written Informed Consent form and be willing to undergo cataract surgery for the bilateral implantation of an intraocular lens (IOL).
* Between the ages of 40 and 80 inclusive on the day the cataract surgery is performed.
* History of Laser-Assisted In Situ Keratomileusis (LASIK), Photorefractive Keratectomy (PRK), Laser-Assisted Subepithelial Keratomileusis (LASEK), Epi-LASIK, or Epi-LASEK more than 1 year prior in both eyes.
* Cataract causing reduction in best corrected distance visual acuity (BCDVA) to a level of 20/40 or worse with or without a glare source in both eyes.
* Willing and able to comply with the requirements for study specific procedures and visits.
* Able to complete a written questionnaire in English.

Exclusion Criteria:

* Prior history of Intacs, RK, CK, AK, Phakic IOL (ICL), Refractive Lens Exchange (RLE), or Corneal Inlay in either eye.
* Pre-existing macular disease in either eye.
* Patients with sufficiently dense cataracts that preclude examination of the macula in either eye.
* History of uveitis in either eye.
* Evidence of ectasia in either eye.
* Previous intraocular surgery in either eye. Eyes with previous pterygium excision are permitted as long as the pterygium did not extend more than 2mm onto the cornea from the limbus.
* Subjects taking systemic medication that may increase sensitivity to UV light.
* Subjects taking a systemic medication that is considered toxic to the retina such as tamoxifen.
* History of ocular herpes simplex virus in either eye.

Ages: 40 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 105 (Actual)
Dates: Start 2018-08-28 (Actual); Primary Completion 2020-04-01 (Actual); Study Completion 2020-04-01 (Actual)

CONTACTS AND LOCATIONS:
Locations (6):
- United States (6):
  - Discover Vision Centers, Leawood, Kansas
  - Cleveland Eye Clinic, Brecksville, Ohio
  - Vance Thompson Vision Clinic, Sioux Falls, South Dakota
  - Slade & Baker Vision, Houston, Texas
  - Focal Point Vision, San Antonio, Texas
  - The Eye Institute of Utah, Salt Lake City, Utah

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Units Other Than Participants: Eyes
Period: Overall Study
Arm/Group | Light Adjustable Lens (LAL) and Light Delivery Device (LDD) | Control IOL
Started | 105; 105 Eyes | 105; 105 Eyes
Completed | 105; 105 Eyes | 105; 105 Eyes
Not Completed | 0; 0 Eyes | 0; 0 Eyes

BASELINE CHARACTERISTICS:
Units Other Than Participants: Eyes
Groups:
- Total: Total of all reporting groups
Arm/Group | Light Adjustable Lens (LAL) and Light Delivery Device (LDD) | Control IOL | Total
Number analyzed (Participants) | 105 | 105 | 210
Number analyzed (Eyes) | 105 | 105 | 210
Age, Continuous [Mean (Standard Deviation); unit: years] | 64.2 (6.9) | 64.2 (6.9) | 64.2 (6.9)
Sex: Female, Male [Count of Units; unit: Eyes]
  Female | 60 | 60 | 120
  Male | 45 | 45 | 90
Ethnicity (NIH/OMB) [Count of Units; unit: Eyes]
  Hispanic or Latino | 12 | 12 | 24
  Not Hispanic or Latino | 93 | 93 | 186
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Units; unit: Eyes]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 0 | 0
  White | 105 | 105 | 210
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Number; unit: Eyes]
  United States | 105 | 105 | 210
Eye [Count of Units; unit: Eyes]
  OD Eye | 52 | 53 | 105
  OS Eye | 53 | 52 | 105

OUTCOME MEASURES:

1. Primary Outcome: Magnitude of Manifest Cylinder (MRCYL) Compared Between the Two Study Groups, LAL and Control
Time Frame: Postop Month 6
Measure: Mean (Standard Deviation); unit: Diopter
Units Other Than Participants: Eyes
Arm/Group | Light Adjustable Lens (LAL) and Light Delivery Device (LDD) | Control IOL
Number analyzed (Participants) | 105 | 105
Number analyzed (Eyes) | 105 | 105
Diopter | -0.319 (0.319) | -0.452 (0.456)

2. Primary Outcome: Absolute Manifest Refraction Spherical Equivalent (MRSE) Compared Between the Two Study Groups, LAL and Control
Time Frame: Postop Month 6
Measure: Mean (Standard Deviation); unit: Diopter
Units Other Than Participants: Eyes
Arm/Group | Light Adjustable Lens (LAL) and Light Delivery Device (LDD) | Control IOL
Number analyzed (Participants) | 105 | 105
Number analyzed (Eyes) | 105 | 105
Diopter | 0.269 (0.269) | 0.379 (0.338)

3. Primary Outcome: One Sided Upper 95% Confidence Limit of the Percentage of LAL Implanted Eyes With BCDVA of 20/40 or Better is Higher Than the Performance Rate of 92.5%
Time Frame: Postop Month 6
Measure: Number (95% Confidence Interval); unit: percent of eyes w. BCDVA 20/40 or better
Units Other Than Participants: Eyes
Arm/Group | Light Adjustable Lens (LAL) and Light Delivery Device (LDD)
Number analyzed (Participants) | 105
Number analyzed (Eyes) | 105
percent of eyes w. BCDVA 20/40 or better | 100 [100 to 100]

4. Secondary Outcome: Uncorrected Distance Visual Acuity (UCDVA)
Time Frame: Postop Month 6
Measure: Mean (Standard Deviation); unit: logMAR
Units Other Than Participants: Eyes
Arm/Group | Light Adjustable Lens (LAL) and Light Delivery Device (LDD) | Control IOL
Number analyzed (Participants) | 105 | 105
Number analyzed (Eyes) | 105 | 105
logMAR | 0.002 (0.108) | 0.052 (0.130)

5. Secondary Outcome: Uncorrected Distance Visual Acuity (UCDVA) for Subjects Measured With Keratometric Cylinder (Kcyl) <0.75 D in Both Eyes at the Preoperative Examination
Time Frame: Postop Month 6
Measure: Mean (Standard Deviation); unit: mean logMAR UCDVA
Units Other Than Participants: Eyes
Arm/Group | Light Adjustable Lens (LAL) and Light Delivery Device (LDD) | Control IOL
Number analyzed (Participants) | 42 | 42
Number analyzed (Eyes) | 42 | 42
mean logMAR UCDVA | -0.003 (0.113) | 0.061 (0.139)

ADVERSE EVENTS:
Time Frame: Through study completion, an average of 6 months
Description: Non-ocular, Non-serious adverse events were not required to be collected per protocol. All-Cause Mortality and Non-Ocular Serious Adverse Events are reported at the participants level. Ocular Serious and Other (Not Including Serious) Adverse Events are presented with total number of eyes monitored/assessed as the at Risk population.
Arm/Group | Light Adjustable Lens (LAL) and Light Delivery Device (LDD) | Control IOL
All-Cause Mortality (participants affected / at risk) | 0/105 | 0/105
Serious Adverse Events (participants affected / at risk) | 1/105 | 0/105
Other Adverse Events (participants affected / at risk) | 48/105 | 38/105
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Light Adjustable Lens (LAL) and Light Delivery Device (LDD) (N=105) | Control IOL (N=105)
Clinically significant Cystoid Macular Edema (Eye disorders) | 0 (0) | 0 (0)
Secondary Surgical Intervention (excluding Posterior Capsulotomy) (Eye disorders) | 1 (1) | 0 (0) — Iris Prolapse secondary to fall requiring Iris Repositioning + Suture
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Light Adjustable Lens (LAL) and Light Delivery Device (LDD) (N=105) | Control IOL (N=105)
Anterior Chamber Inflammation (Eye disorders) | 2 (2) | 2 (2)
Corneal Edema (Eye disorders) | 2 (2) | 0 (0)
Loss of BCDVA of >/= 10 letters (when compared to Preoperative or Postop Week 3 BCDVA) (Eye disorders) | 1 (1) | 0 (0)
Removal of retained Cortex (Eye disorders) | 0 (0) | 1 (1)
Conjunctival hyperemia (Eye disorders) | 1 (1) | 0 (0)
Conjunctival hyperemia/edema (Eye disorders) | 1 (1) | 1 (1)
Corneal SPK (Eye disorders) | 1 (1) | 0 (0)
Double vision (Eye disorders) | 1 (1) | 1 (1)
Epiretinal membrane (Eye disorders) | 0 (0) | 1 (1)
Epithelial basement membrane dystrophy appearance (Eye disorders) | 1 (1) | 0 (0)
Epithelial defect (Eye disorders) | 0 (0) | 2 (2)
Glare at night (Eye disorders) | 0 (0) | 1 (1)
Iris atrophy/Medication deposits (Eye disorders) | 1 (1) | 0 (0)
Iris prolapse (Eye disorders) | 1 (1) | 0 (0)
Light sensitivity (Eye disorders) | 2 (2) | 2 (2)
Non-clinically significant cystoid macular edema (Eye disorders) | 0 (0) | 1 (1)
Ocular discomfort (Eye disorders) | 3 (3) | 1 (1)
Posterior vitreous detachment (Eye disorders) | 0 (0) | 1 (1)
Retained cortex (Eye disorders) | 0 (0) | 1 (1)
Vision doesn't fuse together for distance well (Eye disorders) | 1 (1) | 0 (0)
Vitreous hemorrhage (Eye disorders) | 0 (0) | 1 (1)
Vitreous in anterior chamber (Eye disorders) | 0 (0) | 1 (1)
YAG performed to treat capsular phemosis (Eye disorders) | 1 (1) | 0 (0)
YAG performed to treat capsular striae (Eye disorders) | 1 (1) | 0 (0)
YAG performed to treat posterior capsular opacity (Eye disorders) | 27 (27) | 20 (20)
YAG performed to treat vitreous strand (Eye disorders) | 1 (1) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2019-07-03): https://cdn.clinicaltrials.gov/large-docs/65/NCT03660865/Prot_SAP_000.pdf